CLINICAL TRIAL: NCT05541926
Title: Scaling up eConnect in Juvenile Probation Settings: a Hybrid Implementation Effectiveness Trial of a Digital Suicide Risk/Behavior Identification and linkage-to Treatment System
Brief Title: Scaling up e-Connect in Juvenile Probation Settings
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Indiana University School of Medicine (Other); George Mason University (Other); Chestnut Health Systems (Other); National Institute of Mental Health (NIMH) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Katherine Elkington, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 8359; R01MH130845 (NIH)
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Connect (Experimental): County receives training and materials and subsequently begins the e-Connect intervention
  Interventions: Behavioral: e-Connect
- Standard of Care (No Intervention): Standard of care practice in counties prior to the implementation of e-Connect

INTERVENTIONS:
Behavioral: e-Connect — Implementation of the e-Connect system
  Arms: e-Connect

SUMMARY:
We propose to conduct research on strategies that support the successful scale-up of an evidence-based, suicidal risk and behavior identification and cross-system linkage programs for justice-involved youth (e-Connect), and to rigorously evaluate the implementation activities and associated costs that support that scale-up of e-Connect within 9 Indiana counties. Guided by the GPM and EPIS frameworks, this 4-year study will comprise 3 project phases: (1) Scale-Up Strategy Efforts, focused on preparing for scale-up; (2) e-Connect-scaleup implementation (2a Exploration and Preparation and 2b Implementation and Sustainment); and (3) Scale-Up Effectiveness Trial/Outcome Evaluation. The current project draws on lessons learned from the e-Connect efficacy trial in NYS and research team leadership will serve as External Facilitators to support 9 Local Facilitators to ensure the successful transfer of knowledge, skill and expertise in delivering e-Connect in a new JJ system and geographic context, utilizing implementation strategies to support the more widespread, sustained and rigorous adoption of e-Connect. The study will include a learning community created by External Facilitators for Local Facilitators to provide support, to exchange strategies to handle implementation issues, to develop competencies in facilitation, and to guide implementation throughout the program. The learning community will help Local Facilitators navigate through the implementation stages of the study.

DETAILED DESCRIPTION:
The proposed study will examine strategies to bolster the successful scale-up of e-Connect, one of the few evidence-based suicide behavior identification and cross-system linkage programs for youth on under community supervision. This proposal is from two PIs with complimentary expertise in the justice system, implementation science, clinical decision support systems, and use of large administrative data sets, and is supported by a strong multi-disciplinary team to achieve study aims. Guided by the gateway provider model (GPM) and the Exploration, Preparation, Implementation Sustainment (EPIS) implementation framework, we now propose to extend our work of e-Connect, to develop and test a "purveyor model" of implementation scale-up (i.e. e-Connect-scaleup). In e-Connect-scaleup, research team leadership will serve as External Facilitators to support Local Facilitators to ensure the successful transfer of knowledge, skill and expertise in delivering e-Connect in a new JJ system and geographic context, utilizing implementation strategies to support the more widespread, sustained and rigorous adoption of e-Connect. Working in 9 Indiana counties, randomly assigned to one of three waves in a stepped-wedge, implementation-effectiveness hybrid type-2 design, the specific aims are to examine the clinical and cost-effectiveness of e-Connect-scaleup on (i) identification of youth service need (SB and BH correlates) in juvenile probationers; (ii) cross-system (probation-BH agency) referral; and (iii) youth BH service use (initial BH contact; primary outcome) by comparing the performance of e-Connect to (a) standard probation officer practice (baseline) and (b) to rates achieved in the prior efficacy trial of e-Connect (Aim 1). We will examine potential mediating or moderating effects of EPIS/GPM inner and outer context factors We will also determine whether, at scale, e-Connect promotes SB/BH service need identification, cross-system referral and youth SB/BH service use as compared with standard probation practice (baseline), for all youth on probation, regardless of youth clinical need or demographic characteristics, which would replicate previous performance of e-Connect in NYS (Aim 2). Finally, we will examine the implementation of e-Connect-scaleup in terms of fidelity and acceptability and compare advancement through the stages of implementation through to sustainment across the 9 counties in order to demonstrate the feasibility of scaling-up e-Connect in probation settings beyond NYS (Aim 3). We will elucidate the inner- and outer-level EPIS- and GPM- derived factors that promote or hinder delivery of implementation strategies and practice change to inform scale up across a variety of contexts.

Settings. The sample for the proposed study will be recruited from probation staff, partnering treatment agency staff, and probation youth from 9 counties in Indiana, which are distributed across the state geographically. The counties range in population density, with 5 qualifying as Rural/Mixed and 4 as Urban. Each county participating in the proposed study is also a member of the Indiana Juvenile Detention Alternatives Initiative, a nationwide juvenile justice reform effort funded by the Annie E. Casey Foundation and adopted in nearly a third of Indiana counties. The focus of JDAI is to limit the unnecessary detainment of low-risk probation youth. Each JDAI county has developed committees of staff and community members that use a data-driven process, one of the JDAI core strategies, to identify targets of intervention, assess effectiveness of the interventions, and continue monitoring progress to develop future interventions. Recognizing the benefits of JDAI, Indiana was the second state to institute a central JDAI office to support statewide expansion. Each JDAI county has a dedicated coordinator who will also act as Local Facilitator for e-Connect. See the map indicating the location of participating sites relative to other JDAI counties and juvenile detention centers.

Design, Sample Size and Randomization. In the proposed cluster randomized stepped-wedge design, 9 Indiana counties will be randomized - stratified by population density/urbanicity (as a proxy for staffing and resource availability) - to one of 3 waves of e-Connect-scale-up at 3-month intervals.

We will examine the clinical and cost-effectiveness of e-Connect-scaleup on (i) identification of youth service need (SB and BH correlates) in juvenile probationers; (ii) cross-system (probation-BH agency) referral; and (iii) youth BH service use (initial BH contact; primary outcome) by comparing the performance of e-Connect to (a) standard probation officer practice (baseline) and (b) to rates achieved in the prior efficacy trial of e-Connect (Aim 1). We will examine potential mediating or moderating effects of EPIS/GPM inner (e.g. staff knowledge, organizational functioning) and outer context factors (e.g. youth age, county rate of SB) on e-Connect-scaleup outcomes. We will also determine whether, at scale, e-Connect promotes SB/BH service need identification, cross-system referral and youth SB/BH service use as compared with standard probation practice (baseline), for all youth on probation, regardless of youth clinical need or demographic characteristics, which would replicate previous performance of e-Connect in NYS (Aim 2). Finally, we will evaluate the implementation of e-Connect-scaleup in two ways (Aim 3). First, we will examine the fidelity and acceptability of e-Connect-scaleup, including facilitation strategies. Second, we will document processes of scaling up e-Connect, comparing advancement through the stages of implementation through to sustainment across the 9 counties in order to demonstrate the feasibility of scaling-up e-Connect in probation settings beyond NYS; we will explore the role of site differences and other EPIS and GPM factors on implementation completion (Aim 3). By randomizing sites to e-Connect-scaleup across time, the control group (which is changing over time) is taken to be the sites that have not yet rolled out e-Connect-scaleup by a particular time, treatment as usual (TAU). Data on these behavioral health care cascade outcomes are collected in each county pre and post randomization to e-Connect-scaleup allowing for within site estimates of change while controlling for secular changes over time. We will also examine potential effect modifiers of e-Connect by youth, staff and county level inner and outer setting factors. To examine impact and success of implementation strategies, we will compare stages of implementation completion as well as feasibility and acceptability cross the 9 new counties, exploring the role of site differences as well as other EPIS factors (outer-, inner-context level) on implementation completion. There are two limitations to cluster randomized deigns: potential of uneven distribution of potentially confounding variables within a cluster (i.e. county) as well as interrelationship between variables. Our proposed stratification plan and use of propensity matching will address issues related to confounding. We calculated our ability to detect an effect of e-Connect-scaleup (i.e. power) using a conservative intraclass correlation coefficient (ICC) of .65, denoting a moderate-large positive correlation between outcomes within a county to address issues of interrelationship between variables at the county level.

ELIGIBILITY:
Sample: County Probation Staff

Inclusion Criteria:

* All probation agency leadership and officers employed by the partnering sites who are (a) at least 18 years of age and (b) conversant in English in participating study counties are eligible

Exclusion Criteria:

* There are no exclusionary criteria and no special classes of participants.

Sample: County Treatment Staff

Inclusion Criteria:

* All treatment staff (agency directors, supervisors and clinical line staff) employed by participating treatment agencies who are at least 18 years of age and conversant in English in participating study counties will be asked to participate

Exclusion Criteria:

* There are no exclusionary criteria and no special classes of participants.

Sample: Local Facilitators

Inclusion Criteria:

* All county/local Justice Diversion Alternatives Initiative (JDAI) representatives that work with partnering sites who (a) are at least 18 years of age and (b) conversant in English in participating study counties are eligible

Exclusion Criteria:

* There are no exclusionary criteria and no special classes of participants.

Sample: Probation Youth

Inclusion Criteria:

* All youth who are on probation who are (a) 10-18 years of age and (b) conversant in English in participating study counties are eligible;

Exclusion Criteria:

* There are no exclusionary criteria and no special classes of participants.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3629 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment initiation | 3 years
  Date of first behavioral health appointment/contact; extracted from Indiana Probation management information system (MIS)

SECONDARY OUTCOMES:
Treatment engagement | 3 years
  # of weeks in treatment, via termination date; extracted from MIS, Medicaid data
Screen/Identify Youth Service Need | 3 years
  Via e-Connect system and recorded in Caseload Explorer: YASI Orbis, Chestnut Information indicates whether screening has occurred; Extracted from MIS
Cross-system Referral | 3 years
  Indicated by Referral Date; extracted from MIS
Uptake Adoption of e-Connect system | 6 months
  Acceptability, uptake and sustainability of e-Connect (BH and JJ staff; External and Local facilitators
Uptake Adoption - MIS | 3 years
  Number of eligible youth screened via e-Connect
Fidelity to use of e-Connect system | 3 years
  Measured by Stages of Implementation Completion (SIC) tool. indicated by implementation stages complete; time to stage completion; activities completed w/in each stage)
Fidelity of Facilitation | 3 years
  Checklists (self and observer) documenting completeness of activities; External/Local Facilitation activity tracker
Acceptability of e-Connect by the family | 3 years
  PO completes family debriefing checklist: family receptivity to screening results and referral plan
Sustainability of e-Connect protocol | 1 year, 4 months
  Measured using MIS
Sustainability achieved in implementation process | 1 year, 4 months
  Stages of Implementation Completion (SIC) tool measures - Implementation stages complete; time to stage completion; activities completed within each stage measured by the SIC tool

OTHER OUTCOMES:
Suicidal Behavior, Non-Suicidal Self-Injury (NSSI), BH knowledge | 3 years
  Measured during pre-post quizzes following web-based training modules; developed for study
Perceived importance of screening and referral to BH - Exploration Phase services | 2 months
  Subscales for screening - Measure assessing perceived importance of activities associated with screening, referral and linkage - developed by JJTRIALS research cooperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University and New York State Psychiatric Instititute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No